CLINICAL TRIAL: NCT01529151
Title: Effectiveness of Osteopathic Manipulative Treatment (OMT) and Vestibular Rehabilitation Therapy (VRT) Alone or in Combination on Balance and Visual Function in Individuals With Vertigo and Somatic Dysfunction
Brief Title: Effectiveness of Osteopathic Manipulative Treatment (OMT) and Vestibular Rehabilitation Therapy (VRT) in Individuals With Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 11/IRB/033; 11-13-647 (Other Grant/Funding Number: American Osteopathic Association Council on Research and Osteopathic Heritage Foundation)
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Vertigo; Dizziness; Benign Paroxysmal Positional Vertigo; Labyrinthitis
Keywords: Dizziness; Vertigo; Benign Paroxysmal Positional Vertigo; Labyrinthitis; Osteopathic Manipulative Treatment; Vestibular Rehabilitation Therapy
MeSH Terms: conditions — Vertigo; Dizziness; Benign Paroxysmal Positional Vertigo; Labyrinthitis | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- OMT Group (Active Comparator): Participants will receive Osteopathic Manipulative Treatment (OMT) with the objective of treating diagnosed somatic dysfunction and this will entail the use of specific indirect and direct techniques, including soft tissue, inhibitory, myofascial release, articulatory and high-velocity / low-amplitude (HVLA) techniques.
  Interventions: Other: Osteopathic Manipulative Treatment (OMT)
- VRT Group (Active Comparator): Participants will receive Vestibular Rehabilitation Therapy (VRT), which includes balance exercises in sitting and standing positions that include gaze stabilization, kinesthetic and proprioceptive retraining.
  Interventions: Other: Vestibular Rehabilitation Therapy (VRT)
- OMT - VRT Group (Active Comparator): Participants will receive both Osteopathic Manipulative Treatment (OMT) and Vestibular Rehabilitation Therapy (VRT).
  Interventions: Other: Osteopathic Manipulative Treatment (OMT); Other: Vestibular Rehabilitation Therapy (VRT)
- Control Group (No Intervention)

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment (OMT) — Direct action OMT procedures, including HVLA, involve the application of a force in the direction of restricted joint motion in order to resolve somatic dysfunction. Indirect techniques, including counterstrain, balanced ligamentous tension and myofascial release, entail applying a force away from the restrictive barrier of a joint or soft tissue structure.
  Other Names: Osteopathic Manipulative Medicine (OMM)
  Arms: OMT - VRT Group; OMT Group
Other: Vestibular Rehabilitation Therapy (VRT) — Participants categorized as having a peripheral motion hypersensitivity will receive habituation exercises that reproduce the provocative motion, seated and standing balance exercises with gaze stabilization, kinesthetic and proprioceptive retraining. Participants will be given a monthly exercise log at onset and will be asked to report exercise levels at subsequent follow up periods.
  Arms: OMT - VRT Group; VRT Group

SUMMARY:
Western University of Health Sciences is seeking men and women to participate in a study on the effectiveness of Osteopathic Manipulative Treatment (OMT) and Vestibular Rehabilitation Therapy (VRT) in patients with vertigo. The purpose of this study is to examine the efficacy of OMT in the treatment of individuals with vertigo, alone and in combination with Vestibular Rehabilitation Therapy (VRT). Because of the health care costs associated with vertigo, the cost effectiveness of OMT and VRT will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of dizziness or a diagnosis of vertigo for longer than 3 months duration
* Able to tolerate 30 minutes of sitting and standing
* Able to transfer from sitting to standing and move independently
* Able tolerate manual therapy and exercise

Exclusion Criteria:

* Severe traumatic injury
* Bleeding disorders and anticoagulation (Coumadin) therapy
* Currently receiving VRT, vision therapy, or manual medicine (OMT, Chiropractic, etc.) or received manual medicine within the past three months
* Down syndrome
* Ehlers-Danlos syndrome
* Endolymphatic Hydrops
* Legal blindness in one or both eyes
* Menieres disease
* Neurological conditions (including Peripheral Neuropathy, Stroke, traumatic brain injury, cerebral aneurysm, and Multiple Sclerosis)
* Rheumatoid Arthritis
* Spinal trauma or history of cervical spine surgery

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Dizziness Handicap Inventory (DHI) at 1 week | Baseline to 1 week
  The Dizziness Handicap Inventory (DHI) is a questionnaire that was developed to measure the self-perceived level of handicap associated with the symptom of dizziness.
Change from Baseline in Dizziness Handicap Inventory (DHI) at 3 weeks | Baseline to 3 weeks
  The Dizziness Handicap Inventory (DHI) is a questionnaire that was developed to measure the self-perceived level of handicap associated with the symptom of dizziness.
Change from Baseline in Dizziness Handicap Inventory (DHI) at 12 weeks | Baseline to 12 weeks
  The Dizziness Handicap Inventory (DHI) is a questionnaire that was developed to measure the self-perceived level of handicap associated with the symptom of dizziness.
Change from Baseline in Computerized Dynamic Posturography (CDP) at 1 week | Baseline to 1 week
  Computerized dynamic posturography (CDP), also called test of balance (TOB), is a non-invasive specialized clinical assessment technique used to quantify the central nervous system adaptive mechanisms (sensory, motor and central) involved in the control of posture and balance, both in normal (such as in physical education and sports training) and abnormal conditions (particularly in the diagnosis of balance disorders and in physical therapy and postural re-education).
Change from Baseline in Computerized Dynamic Posturography (CDP) at 3 weeks | Baseline to 3 weeks
  Computerized dynamic posturography (CDP), also called test of balance (TOB), is a non-invasive specialized clinical assessment technique used to quantify the central nervous system adaptive mechanisms (sensory, motor and central) involved in the control of posture and balance, both in normal (such as in physical education and sports training) and abnormal conditions (particularly in the diagnosis of balance disorders and in physical therapy and postural re-education).
Change from Baseline in Computerized Dynamic Posturography (CDP) at 12 weeks | Baseline to 12 weeks
  Computerized dynamic posturography (CDP), also called test of balance (TOB), is a non-invasive specialized clinical assessment technique used to quantify the central nervous system adaptive mechanisms (sensory, motor and central) involved in the control of posture and balance, both in normal (such as in physical education and sports training) and abnormal conditions (particularly in the diagnosis of balance disorders and in physical therapy and postural re-education).

SECONDARY OUTCOMES:
Change from Baseline in Neuro-Optometric Evaluation at 1 week | Baseline to 1 week
  Evaluation of visual acuity and refractive status, oculomotor function and visual field status.
Change from Baseline in Neuro-Optometric Evaluation at 3 weeks | Baseline to 3 weeks
  Evaluation of visual acuity and refractive status, oculomotor function and visual field status.
Change from Baseline in Neuro-Optometric Evaluation at 12 weeks. | Baseline to 12 weeks
  Evaluation of visual acuity and refractive status, oculomotor function and visual field status.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Fraix, DO, Principal Investigator — Western University of Health Sciences
Locations (1):
- Western University Physical Therapy Research Laboratory, Pomona, California, United States

REFERENCES:
- [Background] Fraix M. Osteopathic manipulative treatment and vertigo: a pilot study. PM R. 2010 Jul;2(7):612-8. doi: 10.1016/j.pmrj.2010.04.001. PMID 20659716
- [Derived] Fraix M, Badran S, Graham V, Redman-Bentley D, Hurwitz EL, Quan VL, Yim M, Hudson-McKinney M, Seffinger MA. Osteopathic manipulative treatment in individuals with vertigo and somatic dysfunction: a randomized, controlled, comparative feasibility study. J Osteopath Med. 2021 Jan 1;121(1):71-83. doi: 10.7556/jaoa.2020.147. PMID 33125033